CLINICAL TRIAL: NCT06638944
Title: Impact of Wearable Biofeedback for the Rehabilitation and Tele-rehabilitation of Neurogenic Dysphagia
Brief Title: Wearable Biofeedback for Swallowing Disorders Rehabilitation in Stroke and Parkinson Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Georgia A. Malandraki, Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2024-2; 1R01AG086371-01 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dysphagia; Stroke; Parkinson Disease
Keywords: biofeedback; dysphagia; oropharyngeal dysphagia; Parkinson disease; stroke; telehealth; wearable
MeSH Terms: conditions — Deglutition Disorders; Stroke; Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IN-person i-Phagia (Experimental): The treatment group assigned to the IN-PERSON i-Phagia service delivery will use the system to complete a standardized swallowing rehabilitation protocol for 12 weeks with weekly (once per week) treatment sessions in the clinic and 3 days of home practice per week.
  Interventions: Behavioral: In-person sEMG-biofeedback
- Remote i-Phagia (Active Comparator): The treatment group assigned to the REMOTE i-Phagia service delivery will use the i-Phagia system to complete a standardized swallowing rehabilitation protocol for 12 weeks with weekly (once per week) treatment sessions completed remotely (via telehealth) and 3 days of home practice per week.
  Interventions: Behavioral: Remote sEMG-biofeedback
- Standard-of-Care (SOC) Swallow Treatment (Other): The treatment group assigned to the SOC service delivery will complete the same standardized swallowing rehabilitation protocol and in the same frequency as the i-Phagia groups but without the device. That is, they will complete the protocol for 12 weeks with weekly (once per week) treatment sessions completed in-person and 3 days of home practice per week.
  Interventions: Behavioral: Standard-of-care treatment

INTERVENTIONS:
Behavioral: In-person sEMG-biofeedback — Participants in this intervention complete a standardized behavioral swallowing rehabilitation protocol for 12 weeks with weekly (once per week) treatment sessions in the clinic and 3 days of home practice per week using the i-Phagia sEMG system. The protocol includes oropharyngeal strength training and skill-based practice exercises. For this group, patients use the sensor patch and the software guides them on how to complete the exercises and receive feedback.
  Arms: IN-person i-Phagia
Behavioral: Remote sEMG-biofeedback — Participants in this intervention complete a standardized behavioral swallowing rehabilitation protocol for 12 weeks with weekly (once per week) treatment sessions completed remotely (via telehealth) and 3 days of home practice per week. The protocol includes oropharyngeal strength training and skill-based practice exercises. For this group, patients also use the sensor patch and the software guides them on how to complete the exercises and receive feedback.
  Arms: Remote i-Phagia
Behavioral: Standard-of-care treatment — Participants in this intervention will complete the same standardized behavioral swallowing rehabilitation protocol and in the same frequency as the sEMG biofeedback intervention groups but WITHOUT a device. That is, they will complete the protocol for 12 weeks with weekly (once per week) treatment sessions completed in-person and 3 days of home practice per week. For this intervention group, patients use a visual analog scale and a timer as feedback tools, as frequently done in clinical practice where sEMG devices are not widely available.
  Arms: Standard-of-Care (SOC) Swallow Treatment

SUMMARY:
Dysphagia, or difficulty swallowing, is a common symptom of many neurological diseases but its treatment is not well established or easily accessible.

To start addressing this gap, the researchers developed and validated a cost-effective wearable surface electromyography (sEMG) biofeedback sensor technology (i-Phagia), optimized to record muscle activity from the head/neck and provide biofeedback to patients and adherence data to clinicians during swallow therapy. This system has been developed with commercially available and widely used materials and the Purdue University IRB has determined that the device is non-significant risk device.

The goal of this clinical trial is to learn if this biofeedback (using this new technology/i-Phagia) when used as an adjunct to a standard swallow therapy protocol works to improve swallowing function in patients post chronic stroke or diagnosed with Parkinson's disease. It will also help the investigators learn whether this therapy protocol is equally effective when provided in-person versus via telehealth. Finally, it will determine which patient factors may influence how well the treatment works.

The main questions it aims to answer are:

* Does biofeedback (using this new technology/i-Phagia) when used as an adjunct to a standard swallow therapy protocol works better than a standard of care treatment to improve swallowing function in patients post chronic stroke or diagnosed with Parkinson's disease?
* Is completing the swallow therapy protocol at home (via telehealth) as effective as completing it in-person (in the clinic)?
* What factors related to the patients (e.g., age, diagnosis, etc.) may influence how well the treatment works?

Participants will:

* Complete a 12-week swallow treatment protocol (12 treatment visits) either in-person or at home (via telehealth)
* Complete 3 in-person evaluations (pre-treatment; post-treatment; and at a 12-week post treatment follow-up time point)
* Exercise at home several days per week and keep a diary/log of their home exercise

The hypothesis is that upon study completion, the efficacy of sEMG biofeedback-facilitated swallow therapy for both in-person and telehealth service delivery in two neurogenic dysphagia populations will have been established, and variables determining response to treatment will begin to be identified.

ELIGIBILITY:
Inclusion Criteria:

* 50-90 years old
* a confirmed (by a neurologist/physician) diagnosis of stroke at least 3 months post event, or of PD (Hoehn and Yahr Stages II-IV)
* score in the normal/mild range on the Montreal Cognitive Assessment (MoCA), determined during an in-house screening
* confirmed oropharyngeal dysphagia, as evaluated during the intervention eligibility assessment by a certified and trained Speech Language Pathologist (SLP)
* accuracy of exercise performance; as evaluated during the intervention eligibility assessment by a certified and trained SLP
* independent (or with caregiver support) use of i-Phagia system post pre-intervention training session; as evaluated during the intervention eligibility assessment by a certified and trained SLP

Exclusion Criteria:

* known allergy to barium or known/suspected perforation or obstruction of the gastrointestinal (GI) tract
* recent history of pneumonia (past 6 months)
* head and neck surgery, radiation or trauma
* a score in the moderate-severe range on MoCA (screened during in-house screening)
* other neurological/neuromuscular disorders (e.g., multiple sclerosis, brain tumor, myositis, etc)
* difficulty complying due to neuropsychological dysfunction determined during the in-house screening
* currently enrolled in swallow or speech therapy
* facial hair in the submental (under the chin) area and refusing to shave.
* known allergies relating to the Ten20® Conductive Paste (this is the conductive paste used to help with sensors signal and adherence to the skin) and/or any of the sensor materials (gold/acrylic) that come into contact with the skin
* no oropharyngeal dysphagia; as evaluated during the intervention eligibility assessment by the certified and trained SLP
* inability to perform the prescribed exercises accurately after a maximum of 12 practice trials; as evaluated during the intervention eligibility VFSS assessment by the certified and trained SLP
* inability to use the system accurately post training (for i-Phagia groups); as evaluated during the intervention eligibility assessment by the certified and trained SLP
* inability to safely swallow (without aspiration) at least one consistency; as evaluated during the intervention eligibility assessment by the certified and trained SLP

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale (PAS) | Pre-treatment; up to 1 week post-treatment; and at a 12-week follow-up
  The Penetration Aspiration Scale (PAS) is an 8-point scale, where 1 indicates a completely safe swallow without any penetration or aspiration present, and 8 indicates the most severe degree of aspiration with no attempt to clear the aspirated material. The PAS will be rated by trained investigators blinded to group/arm and time.
Functional Oral Intake Scale (FOIS) | Pre-treatment; up to 1 week post-treatment; and at a 12-week follow-up
  The Functional Oral Intake Scale (FOIS) is a 7-point ordinal scale (1 indicating nothing by mouth-NPO; and 7 indicating eating without restrictions). It will be rated by the evaluating speech-language pathologist/investigator based on patient report of current diet, to assess functional ability for oral intake.
Normalized sEMG amplitude | Pre-treatment; up to 1 week post-treatment; and at a 12-week follow-up
  Normalized surface electromyography (sEMG) amplitude values during standardized swallow tasks and maneuvers will be collected at the evaluation time points. The sEMG data will be analyzed by blinded to group/arm and time investigators using a custom-made EMG analysis Matlab script.

SECONDARY OUTCOMES:
Swallowing-related Quality of Life (SWAL-QOL) | Pre-treatment; up to 1 week post-treatment; and at a 12-week follow-up
  The SWAL-QOL is a 44-item tool/survey consisting of 10 multi-item scales (food selection, burden, mental health, social functioning, fear, eating duration, eating desire, communication, sleep, and fatigue) ranging in score from 0-100. Higher scores indicate better quality of life.
Patient Satisfaction | From date of treatment initiation until the date of the post-treatment evaluation, assessed up to 13 weeks
  Satisfaction and ease-of-use/comfort with the modality (in-person; remote), and materials used (e.g., i-Phagia), will be examined as a secondary variable using a 10-item survey with a positive centered 10-point Likert scale. Possible scores 0-100. Higher values indicate better or higher satisfaction/comfort scores.
Treatment adherence | From date of treatment initiation until the date of the post-treatment evaluation, assessed up to 13 weeks
  Treatment adherence will be calculated as a percent - number of treatment days when all exercises are completed over the total number of treatment days.

OTHER OUTCOMES:
Stimulability | Pre-treatment
  Stimulability is operationally defined as the ability to accurately perform the swallowing maneuvers/exercises immediately or quickly when provided with cues or a model. The number of practice trials required to reach accuracy before treatment is initiated will be recorded, and this number will be used for post-hoc analyses on factors influencing treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Malandraki, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the NIH approved data management and sharing plan, all de-identified demographic, clinical (cognitive, psychological), VFSS, quality of life, satisfaction, safety, treatment adherence and stimulability, and electromyographic data will be shared. All data will be shared in their raw pre-processed format. Respondent identifiers will not be shared. All data will be deidentified prior to receipt by the repository.
  In addition to the subject level data described above, the VFSS and EMG protocol designs and the treatment protocol will be shared as well, to facilitate replication.
  This project will use the Purdue University Research Repository (PURR) to publicly share, archive, and preserve the data. PURR utilizes a web-mediated software platform designed for archiving and sharing of scientific data and meets the standards for ISO 16363 Trusted Digital Repositories. Through PURR, investigators that wish to access the data do not need to be affiliated with Purdue University.
Supporting Information: Study Protocol
Time Frame: The data will be published, archived, and freely available to the public at the time of an associated publication or the end of the performance period, whichever comes first. The repository will provide bit-level preservation activities, representation information, and sustained monitoring by repository managers for a period of at least ten years and longer as needed or when required by policy.
Access Criteria: A. Factors affecting subsequent access, distribution, or reuse of scientific data:
  In order to ensure participant consent for data sharing, IRB paperwork and informed consent documents will include language describing plans for data management and sharing data, describing the motivation for sharing, and explaining that personal identifying information will be removed.
  B. Whether access to scientific data will be controlled:
  Access to data will be freely available, however researchers will be asked to cite the data source in their publications.
  C. Protections for privacy, rights, and confidentiality of human research participants:
  Data will be fully de-identified before being uploaded to PURR. No identifying data will be made available at any time.